CLINICAL TRIAL: NCT06737939
Title: Periprostatic Nerve Block vs. Intravenous Ibuprofen for Pain Management During Transrectal Prostate Biopsy: A Prospective Comparative Study
Brief Title: Periprostatic Nerve Block vs. Intravenous Ibuprofen for Pain Management During Transrectal Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Elzem SEN, Assoc. Prof.Dr, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/51
Record Dates: First submitted 2024-12-10; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Pain, Acute
Keywords: Prostate biopsy; ıv ibuprofen; periprostatic nerve block; visual analog scale
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen group (Experimental): Each patient in Group 1 received 400 mg of IV ibuprofen diluted in 100 mL of solution. The infusion was administered over a 30-minute period to ensure proper absorption and minimize adverse effects.
  Interventions: Other: intravenous ibuprofen
- Periprostatic nerve block (Experimental): Periprostatic Nerve Block (PPNB) using 2% lidocaine was administered for pain relief during the prostate biopsy procedure.
  Interventions: Other: periprostatic nerve block

INTERVENTIONS:
Other: intravenous ibuprofen — A systemic analgesic (NSAID) administered intravenously for pain management during prostate biopsy, without the need for additional invasive interventions.
  Arms: Ibuprofen group
Other: periprostatic nerve block — A local anesthetic injection targeting the periprostatic nerves to provide direct pain relief during the biopsy procedure, considered the gold standard for pain management in prostate biopsies.
  Arms: Periprostatic nerve block

SUMMARY:
This study aimed to compare the efficacy of intravenous ibuprofen with peri-prostatic nerve block in pain control during prostate biopsy and to investigate factors influencing pain scores.

DETAILED DESCRIPTION:
This study aimed to compare the efficacy of intravenous (IV) ibuprofen with periprostatic nerve block (PPNB) in controlling pain during prostate biopsy, a common procedure used to diagnose prostate cancer. The study also aimed to investigate factors influencing pain perception during the procedure, such as prostate-specific antigen (PSA) levels, prostate volume, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

Male gender. Scheduled for a prostate biopsy. Prostate-specific antigen (PSA) levels > 4 ng/mL.

Exclusion Criteria:

Renal failure. Liver failure. Neurological disorders (e.g., dementia, Alzheimer's disease, epilepsy, paraplegia).

Rectal disorders. Previous negative prostate biopsy. Chronic anticoagulant therapy or bleeding diathesis. Severe comorbidities. Psychiatric conditions interfering with consent or compliance.

Ages: 45 Years to 82 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study involves a prostate biopsy, which is a procedure specifically related to the prostate gland, only male participants were included. The prostate is an organ found only in men, making this a male-only study population.
Enrollment: 128 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Before the biopsy, During probe insertion and prostate needle insertion,2 hours and 1 day after the procedure
  Pain Assessment using Visual Analog Scale (VAS),The Visual Analog Scale (VAS) is a tool used to measure subjective characteristics or attitudes that cannot be directly measured. It typically consists of a 10 cm (100 mm) horizontal or vertical line, anchored by two endpoints representing extremes of the sensation being measured.
  Range: Scores range from 0 (minimum) to 10 (maximum). Interpretation: Higher scores indicate a worse outcome (e.g., greater pain intensity or distress).
  Description: Participants mark a point along the line that corresponds to the intensity of their experience. The score is determined by measuring the distance (in centimeters or millimeters) from the lower end of the scale to the participant's mark.

SECONDARY OUTCOMES:
Complications | immediately after the intervention/procedure/surgery
  Complications (such as bleeding, nausea vomiting etc)

CONTACTS AND LOCATIONS:
Overall Officials: Elzem Sen, Assoc Prof, Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep University Hospital, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Derived] Baturu M, Sen E. Periprostatic Nerve Block vs. Intravenous Ibuprofen for Pain Management During Transrectal Prostate Biopsy Procedures: A Prospective Comparative Study. Ann Ital Chir. 2025 Sep 16;97(1):119-125. doi: 10.62713/aic.3938. PMID 41537216